CLINICAL TRIAL: NCT06844461
Title: Quality of Life and Decisional Regret in Patients Affected by Acoustic Neuroma
Acronym: QOL-DR-NEUROMA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: QOL-DR-NEUROMA
Record Dates: First submitted 2025-01-28; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-12

CONDITIONS: Quality of Life Outcomes; Acoustic Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Wait-and-scan cohort: Clinico-radiological follow-up with annual brain MRI to detect increase of volume and size of the tumor
- Surgery cohort: Surgical cohort with tumor excision through any possible approach to lateral skull base

SUMMARY:
Italian translation and validation study of two different questionnaire (VSQOL and DRS) about quality of life in patient with acoustic schwannoma.

ELIGIBILITY:
Inclusion Criteria:

* Patient with sporadic acoustic neuroma in follow-up with wait and scan protocol or treated with microsurgical resection with any approach

Exclusion Criteria:

* Patient with NF2
* Patient previuosly treated with RT in the head and neck district
* Patient with pre-treatment facial palsy ipsi and controlateral
* Patient non native italian speakers
* Patient with major mental illness already existing before the acoustic neuroma diagnosis
* Patient with neurological issues such as chronic migraine or postural instability already existing before the acoustic neuroma diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled at the outpatient clinic of an Otolaryngology and Audiology Unit and Neurosurgery Unit of two third level university hospitals in Northern Italy with acoustic neuroma diagnosis between 01/01/2000 and 31/10/2022.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-20 (Actual); Primary Completion 2025-04-20 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
VSQOL-It | From the surgery to the enrollment time (6 months post-treatment) for surgical group. At baseline at enrollment for wait-and-scan group
  Self evaluation of quality of life in patient diagnosed with sporadic acoustic neuroma. It is composed of 40 questions, of which 37 are built on a Likert scale from 1 to 5, where 1 indicates strong disagreement and 5 indicates strong agreement, and 3 with 3 possible answers. The questions relate to 8 domains: Hearing Problems, Postural Instability and Imbalance, Pain, Discomfort, and Tinnitus, Facial or Ocular Issues, Impact on Physical, Emotional, and Social Well-being, Difficulties with Thinking and Memory, Satisfaction or Regret, Impact on Work Activity.
  The score of questions 1 to 33 is reversed, so that a higher score indicates a favorable health status or better quality of life. The scores for questions 1 to 33 are linearly transformed onto a scale from 0 to 100, where 0 indicates poor quality of life and 100 indicates ideal quality of life. The overall score of the index is calculated as the average of the scores of the first six domains, excluding SatisfactionRegret domain
DRS-It | From the surgery to the enrollment time (6 months post-treatment) for surgical group. At baseline at enrollment for wait-and-scan group
  Decisional regret scale to evaluate any regret about the therapeutic choice both in wait-and-scan cohort and surgical cohort. The score ranges from 0 (no regret) to 100 (complete regret). Patients with more than 25pts are considered to have moderate/high regret

SECONDARY OUTCOMES:
PANQOL | From the surgery to the enrollment time (6 months post-treatment) for surgical group. At baseline at enrollment for wait-and-scan group
  Specific quality of life questionnaire in patient with acoustic neuroma composed of 26 questions built on a Likert scale from 1 to 5, where 1 indicates strong disagreement and 5 indicates strong agreement. The questions relate to 7 domains: Hearing (4 questions), Balance (6 questions), Facial Function (3 questions), Energy (6 questions), Anxiety (4 questions), General Health Status (2 questions), and Pain (1 question).
  The score for each domain is calculated as the average of the responses to the questions assigned to it and is linearly transformed onto a scale from 0 to 100, where 0 indicates poor quality of life and 100 indicates ideal quality of life. The overall score of the scale is calculated as the average of the scores of the individual domains.
DASS-21 Questionnaire | From the surgery to the enrollment time (6 months post-treatment) for surgical group. At baseline at enrollment for wait-and-scan group
  Psychometric self-evaluation of depression, anxiety and stress during the study period. 21 items-questionnaire about depression, anxiety and stress during the study period. Each subscale presents a singular score from 0 to 42. Higher scores corresponds to worse emotional outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Aou Bologna, Bologna, Italy